CLINICAL TRIAL: NCT04522531
Title: Effect of Open Kinetic Chain Shoulder Exercises on Scapulothoracic Muscle Activity on Stable and Unstable Ground
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kübra Canli, Clinical Professor, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Hacettepe Universty
Record Dates: First submitted 2020-08-04; First posted 2020-08-21 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Muscle Weakness; Exercise
MeSH Terms: conditions — Muscle Weakness; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise performed on stabil ground (Experimental): Open cinetic chain shoulder exercise will performed on stabil ground. This exercises will be include PNF (flexion-adduction-external rotation pattern), PNF (flexion-abduction-external rotation pattern), scapular plan abduction, external rotation while keeping shoulder in 45 degree abduction. The weight which used during exercise planned according to individuals body weight: 0-59 kg: 3 kg; 60-69 kg: 4 kg; 70-85 kg: 5Kg. Exercises will be carried out in 3 phases consisting of concantric, isometric and eccentric phases. Each phase will be lasted 3 seconds. The time will be checked by using a metronome.
  Interventions: Other: Open cinetic chain shoulder exercise on unstabil ground

INTERVENTIONS:
Other: Open cinetic chain shoulder exercise on unstabil ground — Open cinetic chain shoulder exercise will be performed on BOSU which provides an unstabil ground. This exercises will be include PNF (flexion-adduction-external rotation pattern), PNF (flexion-abduction-external rotation pattern), scapular plan abduction, external rotation while keeping shoulder in 45 degree abduction. The weight which used during exercise planned according to individuals body weight: 0-59 kg: 3 kg; 60-69 kg: 4 kg; 70-85 kg: 5Kg. Exercises will be carried out in 3 phases consisting of concantric, isometric and eccentric phases. Each phase will be lasted 3 seconds. The time will be checked by using a metronome.

SUMMARY:
Exercises used in shoulder rehabilitation compose of open kinetic chain and closed kinetic chain exercises.The force formed on the trunk and legs is transferred to the shoulder in open and closed kinetic chain exercises before shoulder muscles activation. It was shown that trunk and leg muscle activity changes when they are performed in different ground. But it is unknown how this alteration effect shoulder muscle activity. This will be provide a significance approach due to incremented of shoulder muscle activity is important for shoulder rehabilitation setting. To achieve this aim that is rising of muscle activity, various approach is applied including alteration of ground which individual performed exercise on it. And, it was shown that closed cinetic chain exercise which performed on different ground change shoulder muscle activity. However, it is unknown whether alteration of ground effect shoulder muscle activity or not in open cinetic chain exercise. That's why the aim of this study is to investigate alteration of scapulothoracic shoulder muscle activity in open cinetic chain shoulder exercise which enforced different ground.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy
* Right hand dominant
* Ages between 20-45 years
* To be volunteer participate in the study

Exclusion Criteria:

* Having any shoulder pain in current or in the past
* Any previous surgery
* Pain in any part of the body
* Doing regularly a professional sports
* Neurological disease
* Systemic disease

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-03-20 (Estimated); Primary Completion 2023-08-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Muscle recruitment firing | Change from baseline muscle recruitment firing to in 5 minutes after completion of exercise
  EMG analysis will be performed scapulothoracic muscle including upper trapezius, middle trapezius, lower trapezius and serratus anterior muscle. EMG sensors will be placed for each muscle according to SENIAM guidlines. Maximal voluntary isometric contraction will be performed three times for each muscle according to Kendal. Data will be collected during exercise performance which performed on stabil ground as well as unstabil ground using a BOSU (BOSU, Fitness, LLC, San Diego, CA).

SECONDARY OUTCOMES:
Muscle thickness evaluation | Change from baseline muscle recruitment firing to in 5 minutes after completion of exercise
  Muscle thickness will be analysed including upper trapezius, middle trapezius, lower trapezius and serratus anterior muscle during resting and each exercise performance. For muscle thickness evaluation SHMADZU SDU-1200PRO Diagnostic Ultrasound System (Shimadzu, Japan) device will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe Universty, Ankara, Sıhhıye, Turkey (Türkiye)